CLINICAL TRIAL: NCT05224934
Title: Full-target Ultra-hypofractionated Stereotactic Irradiation Orchestrated With Nodule Boost for Retroperitoneal Sarcoma
Brief Title: Preoperative Ultra-hypofractionated Radiotherapy Followed by Surgery for Retroperitoneal Sarcoma (FUSION-01)
Acronym: FUSION-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principle Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-007744
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Soft Tissue Sarcoma; Retroperitoneal Sarcoma; Radiotherapy Side Effect; Ultra-hypofractionated Radiotherapy; Stereotactic Ablative Radiotherapy
Keywords: stereotactic ablative radiotherapy; hypofractionated radiotherapy; retroperitoneal sarcoma; soft tissue sarcoma; peri-operative complications
MeSH Terms: conditions — Sarcoma; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra-hypofractionated radiotherapy (Experimental): Patients receive ultra-hypo-fractionated radiotherapy with 25Gy to 50Gy in five fractions, followed by surgery done at 1 to 2 months post-RT
  Interventions: Radiation: ultra-hypofractionated radiotherapy

INTERVENTIONS:
Radiation: ultra-hypofractionated radiotherapy — stereotactic ablative radiotherapy with 25 to 50Gy in five fractions given preoperatively

SUMMARY:
To investigate the feasibility and peri-operative complications of preoperative hypo-fractionated radiotherapy followed by surgery for retroperitoneal sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Primary soft tissue sarcoma of retroperitoneal or infra-peritoneal spaces of pelvis
* Sarcoma not originated from bone structure, abdominal or gynecological viscera
* All disease can be included safely within one radiotherapy field
* Absence of extension through the sciatic notch or across the diaphragm
* Histologically proven, excluding the following subtypes: Gastro-intestinal stromal tumors (GIST), rhabdomyosarcoma, PNET or other small round blue cells sarcoma, osteosarcoma or chondrosarcoma, aggressive fibromatosis, sarcomatoid or metastatic carcinoma
* ECOG performance status 0 to 2
* American Society of Anesthesiologist (ASA) score ≤2
* Normal renal function: Calculated Creatinine Clearance ≥50ml/min（by Cockcroft-Gault formula）and functional contralateral kidney by differential renal isotope scan
* Normal bone marrow and hepatic function.
* Contraception was needed for female patients of child-bearing age, or male patients whose partner had child-bearing age
* expected life expectancy longer than 5 years
* Written consent form was given prior to treatment
* Can safely be treated by radiotherapy and surgery

Exclusion Criteria:

* metastatic disease
* Tumor was previously treated by radiotherapy
* Involvement of liver, pancreatic head or duodenum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peri-operative complications | From surgery date up to 7 days later
  The proportion of patients who suffer from

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Ning Lu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided